CLINICAL TRIAL: NCT06719544
Title: A Clinical Study to Evaluate the Effect of Enlicitide on the Pharmacokinetics of Lithium in Healthy Adult Participants
Brief Title: A Study of Lithium and Enlicitide in Healthy Adult Participants (MK-0616-034)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0616-034; MK-0616-034 (Other: MSD)
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — Lithium Carbonate; Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lithium Carbonate (Experimental): On Day 1 of Period 1, a single oral dose of lithium carbonate will be administered.
  Interventions: Drug: lithium carbonate
- Enlicitide with Lithium Carbonate (Experimental): On Day 1 of Period 2, a single oral dose of lithium carbonate will be coadministered with a single oral dose of enlicitide.
  Interventions: Drug: lithium carbonate; Drug: enlicitide

INTERVENTIONS:
Drug: lithium carbonate — Oral capsule
  Other Names: lithium
Drug: enlicitide — Oral tablet
  Other Names: enlicitide decanoate; MK-0616/sodium caprate
  Arms: Enlicitide with Lithium Carbonate

SUMMARY:
Researchers have designed a new study medicine called enlicitide decanoate (MK-0616) as a new way to lower the amount of low-density lipoprotein cholesterol (LDL-C) in a person's blood. Enlicitide decanoate will be called "enlicitide" from this point forward. Lithium (also called lithium carbonate) is a medicine used in bipolar disorder.

Researchers want to learn about lithium when taken at the same time with enlicitide.

They want to:

* Measure a person's blood to find out if the amount of lithium in the blood is the same when lithium is taken alone or with enlicitide
* Learn about the safety of lithium when taken alone or with enlicitide and if people tolerate it

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is medically healthy with no clinically significant medical history
* Is a continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history or presence of clinically significant medical or psychiatric condition or disease
* Has a history of cancer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) for Lithium in Plasma | At designated timepoints (up to approximately 5 days post dose)
  Blood samples will be collected to determine the AUC0-inf of lithium in plasma.
Area Under the Concentration versus Time Curve From Time Zero to Last Quantifiable Sample (AUC0-last) for Lithium in Plasma | At designated timepoints (up to approximately 5 days post dose)
  Blood samples will be collected to determine the AUC0-last of lithium in plasma.
Cmax (Maximum Concentration) for Lithium in Plasma | At designated timepoints (up to approximately 5 days post dose)
  Blood samples will be collected determine the Cmax of lithium in plasma.

SECONDARY OUTCOMES:
Number of Participants who experience a Treatment Emergent Adverse Event (TEAE) | Up to approximately 3 weeks
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE will be considered treatment-emergent if the onset date and time is at the time of or after the first study drug administration. The number of participants who experience a TEAE will be reported.
Number of Participants Who Discontinue Study Due to a TEAE | Up to approximately 3 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE will be considered treatment-emergent if the onset date and time is at the time of or after the first study drug administration. The number of participants who discontinue study due to a TEAE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion ( Site 0002), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com